CLINICAL TRIAL: NCT04545983
Title: Long-term Follow-up of Movement of the Cervical Spine After Anterior Cervical Discectomy (ACD) or Anterior Cervical Discectomy With Arthroplasty (ACDA)
Brief Title: Long-term Follow-up Motion Analysis of ACD Versus ACDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zuyderland Medisch Centrum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Z2020101
Record Dates: First submitted 2020-07-28; First posted 2020-09-11 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2021-05

CONDITIONS: Cervical Myelopathy; Cervical Radiculopathy; Spinal Stenosis; Spinal Disease; Spine Degeneration; Spine Fusion
Keywords: Anterior Cervical Discectomy; Anterior Cervical Discectomy with Arthroplasty; ACD; ACDA; Cervical Motion; Long-term Follow-up; Motion Analysis
MeSH Terms: conditions — Radiculopathy; Spinal Stenosis; Spinal Diseases

STUDY DESIGN:
Intervention Model Description: This is a fundamental research project in which a cohort of previously operated patients will be included. All of these patients were previously operated in the setting of an RCT an underwent ACD or ACDA for CDDD. In the RCT flexion and extension cinematographic recordings of the cervical spine were made before surgery, and at three months and one-year post-operatively.
  This study investigates the long-term follow-up of this same study population. The average follow-up duration is 9 years (range 6-13 years). We make similar flexion and extension cinematographic recordings to assess the sequence of segmental contributions of the lower cervical spine years after ACD and ACDA surgery for CDDD. The sROM and level of degeneration will be assessed as a secondary outcome. Moreover, the long-term clinical outcomes will be assessed through questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACD (Active Comparator): In the previously conducted RCT 27 adult patients with an indication for ACD because of a monoradicular syndrome, corresponding to the C5-C6 or C6-C7 level, with corresponding pathology on MRI, were included and randomized to undergo ACD or ACDA.
  Interventions: Other: Motion Analysis
- ACDA (Experimental): In the previously conducted RCT 27 adult patients with an indication for ACD because of a monoradicular syndrome, corresponding to the C5-C6 or C6-C7 level, with corresponding pathology on MRI, were included and randomized to undergo ACD or ACDA.
  Interventions: Other: Motion Analysis

INTERVENTIONS:
Other: Motion Analysis — Cinematographic recordings will be made. Participants are seated on a crutch, adjustable in height, with their neck, shoulders and head free. Before recordings are made, participants will be instructed to perform the prescribed flexion and extension movement in about 10 seconds with 7 frames per second. Participants are placed on the crutch with their shoulder's perpendicular to the image intensifier to obtain sagittal images from the occiput till C7. As soon as the recording is started, the participant is instructed to move his head in the sagittal plane from maximal extension to maximal flexion, without moving the upper part of the body. It is important that the participants shoulders are kept as low as possible while making the recordings to ensure that all the cervical vertebrae are visible. The movement of the cervical spine should be as fluent as possible to prevent for sudden large rotations and translations between consecutive frames.

SUMMARY:
Rationale: Cervical degenerative disc disease (CDDD) is a common cause of cervical radiculopathy, myelopathy or myeloradiculopathy. Surgical treatment is indicated when conservative therapies do not provide sufficient relief or when neurological complaints are progressive. The main surgical techniques are anterior cervical discectomy with (ACDF) or without fusion (ACD), whereas both techniques result in high fusion rates. Short term outcomes of surgery show good clinical results. Long term follow-up shows a drop-in satisfaction rates, often due to the occurrence of new complaints. Pathology is often located at levels adjacent to the previously operated segment, known as adjacent segment disease (ASDis). This is thought to be the results of loss of motion at the previously operated and fused segment. Anterior cervical discectomy with arthroplasty (ACDA) is developed in an effort to reduce the incidence of ASDis by preserving physiological motion in the operated segment.

Objective: To investigate physiological motion of the cervical spine the investigators will analyze motion patterns at the long-term in patients who underwent surgical treatment for CDDD, either ACD or ACDA.

Study design: Fundamental research. This is a prospective study that includes a cohort of patients previously operated in the setting of a randomized controlled trial.

Study population: Adult patients with an indication of surgical treatment for cervical radiculopathy as a consequence of CDDD were enrolled in an RCT between 2007 and 2014 and assigned to undergo ACD or ACDA. Flexion and extension cinematographic recordings of the cervical spine were performed, with the last one at one-year follow-up. The majority of patients in the ACDA group (80%) showed a normal sequence of segmental contribution, which was not the case in the ACD group. This cohort will now be asked to participate in the long-term follow-up study assessing the motion patterns 6-13 years after ACD or ACDA surgery.

Intervention: One flexion and extension cinematographic recording of the cervical spine and will be made.

Main study parameters/endpoints:

The sequence of segmental contributions in sagittal rotation during flexion and extension of the cervical spine will be assessed in the long-term follow-up of surgical treatment. Secondary outcomes will be to assess the amount of degeneration based on the Kellgren Score (KS) and the segmental range of motion (sROM). Long term clinical outcomes will be assessed according to VAS, NDI, SF-36 and Odom's criteria. Patients will be asked whether they have new neurological symptoms and whether they have had a re-operation.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Participants receive cinematographic recordings once. The amount of radiation is a negligible risk. There will be no health benefits. There will be no follow-up.

DETAILED DESCRIPTION:
Cervical degenerative disc disease (CDDD) results from degeneration of cervical intervertebral disc(s) and/or the adjoining vertebral bodies. This causes clinical symptoms of cervical myelopathy, radiculopathy or myeloradiculopathy. Surgical treatment can be an option if non-surgical treatment options provide insufficient relief. The standard surgical technique for treating single or multilevel CDDD is anterior cervical discectomy, either without (ACD) or with fusion (ACDF). Both ACD and ACDF have good short-term clinical results in 90-100% of patients. Both techniques also have a high rate of fusion, respectively 70-80% and 95-100% 1. After 7-20 years, patient satisfaction slowly drops to 68-96% 2. The reason for this decline is thought to be due to the development of adjacent segment disease (ASDis). This is defined as the development of new complaints of radiculopathy or myelopathy due to degeneration one level above or below the previously operated segment. This occurs in approximately 25% of patients during 10 years follow-up and more than 2/3 of these patients need additional surgery 3. The underlying mechanism is thought to be compensation of loss of motion in the fused segment, resulting in overstraining of the adjacent segments 4. Anterior cervical discectomy with arthroplasty (ACDA) is developed in an effort to reduce the incidence of ASDis by preserving physiological motion in the operated segment.

Although the term 'physiological motion' is commonly used, a proper definition has been lacking for a long time. Segmental range of motion (sROM, e.g. the amount of sagittal rotation in a segment between maximal flexion and maximal extension position of the entire cervical spine) is most commonly used to study motion. SROM, however, suffers from large intra- and interindividual variability 5,6. Therefore, in the lower cervical spine, Boselie et al have recently described a consistent sequence of segmental contribution in sagittal rotation during flexion and extension in 80-90% of 20 healthy participants7,8. The normal sequence of segmental contributions in the lower cervical spine during the second half of extension was C4-C5 followed by C5-C6, and then C6-C7.

Moreover, Boselie et al performed a randomized controlled trial (RCT) to compare the presence of this physiological motion pattern and clinical outcomes for ACDA (n=12) and ACD (n=12) patients. Before the randomization 3 patients were operated in a pilot group (all with ACDA), so in total 27 patients with CDDD and radiculopathy were operated. In both groups 10 patients were available for follow-up at one year and fusion rate was 0% in the ACDA group and 70% in the ACD group. The majority of patients in the ACDA group (80%) showed a normal sequence of segmental contribution, which was not the case in the ACD group. This is the first method described which can reliably differentiate between normal or abnormal movement of the cervical spine in an individual subject. There were no differences in patient reported outcome measures, however the study population was small. These data have been submitted but not been published yet since follow-up duration is considered too short for most journals. The primary goal when performing the study was to analyze the sequence of segmental contribution of motion for which a follow-up duration of one year seemed appropriate. However, the expected advantage of the ACDA lies in the long-term, since it should lead to less ASDis by preserving physiological motion in the operated segment. Therefore, longer follow-up is needed to be able to determine if this physiological motion pattern remains present in the ACDA group at the long term. In the RCT performed by Boselie et al, the first patient was operated in December 2007 and the last patient in September 2014. At this moment the follow-up duration is therefore 6 to almost 13 years. By using the same method for analyzing the sequence of segmental contribution of motion in the cervical spine 8, the investigators want to analyze these 27 patients again in the long-term (at an average follow up of 9 years).

The investigators hypothesize that normal motion of the cervical spine will also be preserved by ACDA at the long-term, whereas ACD shows a decline in motion due to the induced fusion at the operated segment. As a consequence, the investigators expect ACDA to induce a lower risk on developing ASDis and thus re-operations.

ELIGIBILITY:
Inclusion criteria for the previous RCT were:

* An indication for ACD because of a monoradicular syndrome, corresponding to the C5-C6 or C6-C7 level, with corresponding pathology on MRI.
* Aged 18-55 years.
* Able to actively perform flexion/extension movement.
* Able to read the information form and sign IC.

For this long-term follow-up study, inclusion criteria are:

* All participants of previous RCT
* Able to perform flexion/extension movement of the cervical spine
* Signed IC.

Patients were excluded in the previous RCT based on the following criteria, and will now be excluded based on the same criteria:

* Ongoing or active infection.
* Previous or actual tumorous processes in the cervical region.
* Pregnancy.
* Previous radiation therapy in the cervical region.
* Not being able to speak Dutch.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-12 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-10-25 (Actual)

PRIMARY OUTCOMES:
Motion Analysis | 9,5 years average
  The sequence of segmental contributions in sagittal rotation during flexion and extension in the lower cervical spine at the long-term after ACDA or ACD surgery for CDDD will be defined. There will be differentiated between normal or abnormal movement amongst ACD and ACDA.
Level of Degeneration | 9,5 years average
  At the start of the cinematographic recording, one image will be saved as a lateral X-ray of the cervical spine to determine Kellgren's Score (KS).
  The KS will be determined by two neurosurgeons and is a scoring method to determine severity of degenerative disc disease, using five gradations:
  * Grade 0: absence of degeneration in the disc.
  * Grade 1: minimal anterior osteophytosis.
  * Grade 2: definite anterior osteophytosis, possible narrowing of the disc space, some sclerosis of the vertebral plates.
  * Grade 3: moderate narrowing of the disc space, sclerosis of the vertebral plates, osteophytosis.
  * Grade 4: severe narrowing of the disc space, severe sclerosis of the vertebral plates, multiple large osteophytes.

SECONDARY OUTCOMES:
VAS Score | 9,5 years average
  Patients will be asked to indicate the VAS score for neck and arm pain (both left and right) will be asked
NDI | 9,5 years average
  The NDI is a modification of the Oswestry Low Back Pain Disability Index. It is a patient- completed, condition-specific functional status questionnaire with 10 items including pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Each section is scored on a 0 to 5 rating scale, in which zero means 'No pain' and 5 means 'Worst imaginable pain'. Al the points can be summed to a total score. The test can be interpreted as a raw score, with a maximum score of 50, or as a percentage. 0 points or 0% means: no activity limitations, 50 points or 100% means complete activity limitation.
SF-36 | 9,5 years average
  The SF-36 health survey will be used to assess both mental and physical health from the patient's perspective
Odom's Outcome Criteria | 9,5 years average
  The Odom's Outcome Criteria will be evaluated in all patients. This score was developed to assess clinical outcomes of cervical degenerative disc surgery
New complaints and/or surgeries | 9,5 years average
  Patients will be asked whether they have new complaints of radiculopathy, myelopathy or myeloradiculopathy and whether they underwent a re-operation for these complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Henk Van Santbrink, Md, PhD, Professor, Principal Investigator — Zuyderland Medisch Centrum
Locations (1):
- Zuyderland Medisch Centrum, Heerlen, Limburg, Netherlands